CLINICAL TRIAL: NCT06027255
Title: Long COVID Immune Profiling
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Cyndya Shibao, MD, Associate Professor, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Long COVID
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Long COVID; POTS - Postural Orthostatic Tachycardia Syndrome; Autonomic Dysfunction
Keywords: SARS-CoV-2 infection; POTS; Orthostatic Intolerance; Long COVID; Long hauler COVID infection
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Postural Orthostatic Tachycardia Syndrome; Primary Dysautonomias; COVID-19; Orthostatic Intolerance

STUDY DESIGN:
Intervention Model Description: To enroll up to 150 patients, 50 POTS without Long-COVID, 50 POTS with Long-COVID and 50 controls with history of COVID-19 infection without sequelae
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Post- COVID 19 POTS patients (Other): Inflammatory markers IL-6,Cytokines (IL-17, and IFN-ɣ), Autonomic symptoms assessment questionnaire (COMPASS 31): In post-COVID-19 POTS (cases).
  Interventions: Diagnostic Test: IL-6; Diagnostic Test: cytokines (IL-17, and IFN-ɣ); Behavioral: Compass 31
- POTS patients (Other): Inflammatory markers IL-6,Cytokines (IL-17, and IFN-ɣ), Autonomic symptoms assessment questionnaire (COMPASS 31):Gender, age, and BMI-matched: patients with diagnosis of POTS
  Interventions: Diagnostic Test: IL-6; Diagnostic Test: cytokines (IL-17, and IFN-ɣ); Behavioral: Compass 31
- Post- COVID 19 POTS patients with Controls (Other): Inflammatory markers IL-6,Cytokines (IL-17, and IFN-ɣ), Autonomic symptoms assessment questionnaire (COMPASS 31):Gender, age, and BMI-matched: Controls are :COVID-19 infected without sequelae
  Interventions: Diagnostic Test: IL-6; Diagnostic Test: cytokines (IL-17, and IFN-ɣ); Behavioral: Compass 31

INTERVENTIONS:
Diagnostic Test: IL-6 — Compare IL-6 level , as a marker of inflammation in all the 3 groups:
  * POTS patients
  * post-COVID-19 POTS
  * gender, age, and BMI-matched controls, with history of COVID-19 infection without sequelae.
Diagnostic Test: cytokines (IL-17, and IFN-ɣ) — Compare Proinflammatory cells and its secreted cytokines (IL-17, and IFN-ɣ) in all the 3 groups:
  * POTS patients
  * post-COVID-19 POTS
  * gender, age, and BMI-matched controls, with history of COVID-19 infection without sequelae
Behavioral: Compass 31 — Autonomic symptoms assessment questionnaire (COMPASS 31), in post-COVID-19 POTS and compare with POTS patients

SUMMARY:
Parasympathetic nervous system (PNS) is part of the body's autonomic nervous system(PNS) protects body against inflammation. Study shows that reduced PNS function activity is associated with persistent inflammation.

Preliminary data from the studies shows, that post-COVID-19 POTS patients have reduced parasympathetic (PNS) function. Given that the PNS protects against inflammation, this clinical trial aims to prove that post-COVID-19 POTS is caused by reduced PNS activity, which in turn, contributes to persistent inflammation, orthostatic intolerance, and OI symptoms.

The study will evaluate immune cell activation in post-COVID-19 POTS and patients with history of COVID-19 infection without sequelae and correlate this with the degree of decreased PNS activity.

DETAILED DESCRIPTION:
COVID-19 infections can cause a disabling syndrome that persists beyond the 3-month convalescence period. The term post-acute COVID-19 syndrome or Long COVID is coined to describe a cluster of symptoms consisting of fatigue, chest pain, reduced exercise tolerance, tachycardia, and cognitive impairment.

Persistent tachycardia remains one of the most common complaints, reported in 9% of patients at 6 months post-infection. These symptoms overlap with those present in patients with Postural orthostatic tachycardia syndrome (POTS). It is noteworthy that about half of POTS patients also report a history of viral infection prior to the development of these symptoms.

Post-COVID-19 tachycardia syndrome, POTS variant: It present with chronic tachycardia with symptoms of orthostatic intolerance (OI) without any other identifiable cause. In addition, non-specific symptoms such as fatigue, headache, and "brain fog", commonly described in POTS patients are also present in this novel condition.

Elevated levels of inflammatory markers CRP,D-dimer and IL-6 are found in Long COVID patients. Data in POTS, which resembles post-COVID tachycardia syndrome, shows increased cytokines including IL-6, IL-1b, and TNF-a.

Notably, stimulation of the efferent vagus nerve (PNS), has been shown to reduce proinflammatory markers production and systemic inflammation. Hence, decreased PNS function, as reported with acute SARS-CoV-2 infection and in post-COVID-19 POTS patients, may render these patients prone to persistent inflammation. To determine the link between PNS activity and immune activation in post-COVID-19 POTS, the study aims to evaluate immune cell activation in post-COVID-19 POTS and patients with history of COVID-19 infection without sequelae and correlate this with the degree of decreased PNS activity.

Rationale and Specific Aims:

Preliminary data shows that post-COVID-19 POTS patients have reduced parasympathetic (PNS) function. Given that the PNS protects against inflammation, we hypothesize that post-COVID-19 POTS is caused by reduced PNS activity, which in turn, contributes to persistent inflammation, orthostatic intolerance, and OI symptoms.

Primary Aim: Test the hypothesis that reduced PNS activity is associated with persistent inflammation in patients with post-COVID-19 POTS.

Study Participants:

This is a cross-sectional study conducted, up to 150 patients will be enrolled, 50 POTS without Long-COVID, 50 POTS with Long-COVID and 50 controls with history of COVID-19 infection without sequelae.

Study Procedures

Recruitment: Subjects will be recruited from referrals to the Vanderbilt Autonomic Dysfunction Center (ADC)

Study visit:

Assessments:

* Autonomic symptoms assessment questionnaire (COMPASS-31)
* Quality of life EQ-5D
* PROMIS scale (Functional Activities Questionnaire in Older Adults with Dementia),
* OHQ (Orthostatic Hypotension Questionnaire)
* CBS (Cambridge Brain sciences: Web based cognitive assessment platform, Optional), and neuropsychological tests Blood sample collection: CBC, CMP, C-reactive protein (CRP), D-dimer, Flow cytometry study, PBMC isolation Autonomic function tests: Testing performed at Vanderbilt ADC within 10 years of the study visit will be utilized. Testing will not be repeated solely for the purposes of this study.

Statistical Considerations

Biostatistical Section The primary endpoint serum IL-6. The proposed sample size of 150 (50 POTD, 50 Long COVID POTS patients and 50 controls) provides more than 90% power to detect an effect size of 0.62 for the mean difference in IL-6 between post-COVID-19 POTS (cases) and controls (COVID-19 infected w/o sequelae), with the two-sided type I error = 5%. This calculation is based on the preliminary data of mean difference of IL-6 ≈ 1.82 and the SD ≈ 2.94 in POTS.16 The effect size is defined as the ratio of mean IL-6 difference between cases and controls to standard deviation.

Data analysis plan: Demographic information will be tabulated. Descriptive statistics, including means, standard deviations, and ranges for continuous parameters, as well as percent and frequencies for categorical parameters, will be presented. T-test or Mann-Whitney (as appropriate) will be applied to examine the mean differences between cases and control with respect to the outcomes. The conditional logistic regression model will be applied for the multivariable data analysis. The adjusted p-values and the adjusted 95% confidence intervals (CIs) will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be 18 years or older, men and women.
* History of confirmed COVID-19 infection (positive contact and symptoms, antigen test or PCR).
* POTS will be defined as the presence of orthostatic tachycardia (>30 bpm) and chronic (>3 months) pre-syncopal symptoms.
* Post-COVID-19 POTS will be defined as the presence of orthostatic tachycardia (>30 bpm) and chronic (>3 months) pre-syncopal symptoms. Symptoms occurred within 2 months after COVID infection and persistent until enrollment in the study.

Exclusion Criteria:

* Individuals with a history of physician diagnosed myocardial infarction, angina, heart failure, stroke, or transient ischemic attack, or who had undergone an invasive procedure for CVD (coronary artery bypass graft, angioplasty, valve replacement, pacemaker placement or other vascular surgeries).
* Inability to comply with the protocol, e.g. uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study.
* Chronic use of steroids, anti-IL6 (omalizumab), anti-TNF-alpha, other immunosuppressants.
* Chronic use of NSAID. Should not enroll if taking without one week prior to blood sampling.
* Treatment with plasmapheresis, IVIG or other immune modulator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
IL-6 levels | Baseline
  Parasympathetic (PNS) function, protects against inflammation. To Evaluate level of inflammation in post-COVID-19 POTS and patients with history of COVID-19 infection without sequelae and correlate this with the degree of decreased PNS activity.
  The primary endpoint is IL-6 levels

SECONDARY OUTCOMES:
Orthostatic Symptoms Score | Baseline
  Standardized Orthostatic Symptoms Score COMPASS-31: Composite Autonomic Symptom Score The COMPASS-31 is a widely-utilized patient questionnaire that provides a quantitative assessment of the severity and distribution of autonomic symptoms . This questionnaire generates a weighted score from 0 to 100, and questions fall into one of six domains: orthostatic intolerance, vasomotor, secretomotor, gastrointestinal, bladder, and pupillomotor function.
cytokines (IL-17, and IFN-ɣ) | Baseline
  Proinflammatory cells and its secreted cytokines (IL-17, and IFN-ɣ) in Post-COVID-19 POTS patients, comparing to controls

CONTACTS AND LOCATIONS:
Locations (1):
- Cyndya Shibao, Nashville, Tennessee, United States